CLINICAL TRIAL: NCT02096237
Title: First in Man Trial to Investigate Safety and Efficacy of the New IgE Adsorber
Brief Title: Extracorporeal SPecific IgE Removal From the Plasma of Allergic Asthma Patients (ESPIRA-study)
Acronym: ESPIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TA-IgE-01-A
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Asthma
Keywords: asthma, bronchial; immunoadsorbents; apheresis; immunoglobulin E
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- apheresis, IgE adsorber (Experimental): 9 apheresis treatments with the new IgE adsorber in a period of 3 months with 3 cycles of 3 treatments each every month.
  Interventions: Device: IgE adsorber
- Conventional drug treatment (No Intervention): Patients treated with conventional asthma treatment as prescribed before study entry. No intervention in prescription

INTERVENTIONS:
Device: IgE adsorber — Two plasma volumes of each patient in the apheresis group will be treated per session
  Arms: apheresis, IgE adsorber

SUMMARY:
In this study patients suffering from Immunoglobulin E (IgE) mediated asthma are treated with a method, called immune apheresis, that removes IgE from blood. In order to achieve this blood is taken continuously from the patient and then separated into plasma and blood cells by centrifuge. The plasma passes the new IgE adsorber where the IgE is specifically bound. The "cleaned" plasma re-joined with the blood cells is given back to the patient. In total each patient randomized to the apheresis group will undergo 3 treatments per week (i.e. 1 cycle) every 4 weeks over a time period of 3 months, that means 9 apheresis treatments in 3 cycles in total. Study hypothesis is that the new IgE adsorber is capable of reducing IgE in plasma/serum by at least 50% measured before the first treatment in the first cycle and after the last treatment in the last treatment cycle. The new adsorber can be safely used in patients. A group of patients with conventional drug treatment and no apheresis treatment serves as control.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Clinically relevant allergy to respiratory allergens confirmed by patient's history, skin-prick testing, IgE serology
* Allergic asthma (diagnosed by lung specialist)
* IgE concentration in blood at least 300 kilo Units (kU)/L

Exclusion Criteria:

* Participation in another trial within 30 days prior to enrolment
* Gravidity (pregnancy test prior to each treatment cycle)
* Intake of omalizumab
* Hepatitis or HIV or malignant disease
* Specific immunotherapy in the last 6 months
* Non-allergic asthma
* Auto-immune diseases
* Hypocalcaemia
* Intake of ACE-inhibitors (discontinuation according to half-time before treatment possible)
* Uncontrolled bleeding and coagulation disorders
* Severe cardiovascular disease
* Severe cardiac arrhythmias
* Severe systemic infection
* Unability to tolerate therapeutic apheresis procedures (hypersensitivity associated with previous apheresis sessions)
* Inadequate peripheral venous access
* Condition in which acute fluid shifts may cause congestive heart failure
* Established or suspected intra-cranial disease where fluid imbalance or pressure changes could exacerbate the disease
* Impaired renal function
* Clinically significant hypotension or borderline hypotension where a further drop in blood pressure could be harmful

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Reduction of IgE concentration in Plasma/Serum | Before first treatment (baseline) to after the last of 9 treatments over a time period of 3 months
  Decrease in IgE concentrations from before the first apheresis treatment (in the control group the first blood sampling) to after the last apheresis treatment after three months (in the control group last blood sampling after three months)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Derfler, Prof. Dr., Principal Investigator — Dep. of Internal Medicine III, Nephrology and Dialysis
Locations (1):
- Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Lupinek C, Derfler K, Lee S, Prikoszovich T, Movadat O, Wollmann E, Cornelius C, Weber M, Froschl R, Selb R, Blatt K, Smiljkovic D, Schoder V, Cervenka R, Plaichner T, Stegfellner G, Huber H, Henning R, Kozik-Jaromin J, Perkmann T, Niederberger V, Petkov V, Valent P, Gauly A, Leinenbach HP, Uhlenbusch-Koerwer I, Valenta R. Extracorporeal IgE Immunoadsorption in Allergic Asthma: Safety and Efficacy. EBioMedicine. 2017 Mar;17:119-133. doi: 10.1016/j.ebiom.2017.02.007. Epub 2017 Feb 12. PMID 28254561